CLINICAL TRIAL: NCT00859781
Title: A Randomized Phase 2 Trial of 177Lu Radiolabeled Monoclonal Antibody HuJ591 (177Lu-J591) and Ketoconazole in Patients With High-Risk Castrate Biochemically Relapsed Prostate Cancer After Local Therapy
Brief Title: 177Lu Radiolabeled Monoclonal Antibody HuJ591 (177Lu-J591) and Ketoconazole in Patients With Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0810010067; J591+Ketoconazole (Other: Weill Cornell Medicine)
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Results first posted 2023-07-19 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — J591 monoclonal antibody; Ketoconazole; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1. 177Lu-J591 + Ketoconazole (Experimental): Ketoconazole 400 mg 3 times a day plus hydrocortisone 20 mg AM, 10 mg PM x 4 weeks followed by 177Lu-J591 Infusion, continue ketoconazole and hydrocortisone
  Interventions: Drug: 177Lu-J591; Drug: Ketoconazole; Drug: Hydrocortisone
- 2. 111In-J591 + Ketoconazole (Placebo Comparator): Ketoconazole 400 mg 3 times a day plus hydrocortisone 20 mg AM, 10 mg PM x 4 weeks followed by 111In-J591 (placebo) Infusion, continue ketoconazole and hydrocortisone
  Interventions: Drug: Ketoconazole; Drug: Hydrocortisone; Drug: 111In-J591

INTERVENTIONS:
Drug: 177Lu-J591 — 177Lu-J591 70 mCi/m2 on day 29 (+/- 2 days) of treatment
  Other Names: J591
  Arms: 1. 177Lu-J591 + Ketoconazole
Drug: Ketoconazole — Ketoconazole at a dose of 400 mg (two 200 mg tabs) to be taken orally (preferably on an empty stomach) three times per day (total daily dose of 1200 mg)
  Other Names: Nizoral
Drug: Hydrocortisone — Hydrocortisone at a dose of 20 mg orally each morning, 10 mg orally each evening (total daily dose of 30 mg)
  Other Names: Cortef
Drug: 111In-J591 — 111In-J591 at a dose of 5 mCi on day 29 (+/- 2 days) of treatment
  Other Names: J591
  Arms: 2. 111In-J591 + Ketoconazole

SUMMARY:
The purpose of this study is to test the effectiveness of the experimental drug, 177Lu-J591 in combination with ketoconazole and hydrocortisone against prostate cancer.

DETAILED DESCRIPTION:
This research is being done because the standard treatments for prostate cancer that has returned (PSA is elevated) after surgery and/or radiation and progressed on initial hormonal therapy are not curative. Existing treatments, such as the ketoconazole used as part of this study may decrease PSA temporarily, but unfortunately the cancer continues to grow. This experimental drug is designed to seek out all of the prostate cancer cells and to deliver a lethal dose of radiation to the areas of cancer, but not to normal areas. Some of the normal organs (liver, kidney and bone marrow) do receive some radiation dose that is within the acceptable limits.

The experimental drug in this study includes an antibody (abbreviated: mAb) called "J591". It is a protein molecule which can bind to a specific site on a prostate cancer cell. A very energetic radioactive (an unstable atom) metal called 177Lutetium (abbreviated: 177Lu) is attached to the J591 antibody. The fully assembled drug is called "177Lu-J591". The study will assess the potential of the energy given off by the radioactive compound to kill cancer cell. This study may also involve the use of 111Indium (abbreviated 111In). This is also an energetic radioactive particle, but does not generally give off enough energy to kill cancer cells, but allows researchers to take pictures. This radioactive particle is also attached to the J591 antibody (called 111In-J591) and will serve as a placebo (treatment with no active medicine).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate previously treated with surgery and/or radiotherapy.
* Biochemical progression (rising PSA) after medical or surgical castration
* High risk of systemic progression defined as:

  1. Rising PSA as defined above and either:
  2. Absolute PSA > 20 ng/mL AND/OR
  3. PSA doubling time < 8 months
* No evidence of local recurrence or distant metastases
* Age >18 years.
* Serum testosterone < 50 ng/ml
* Patients capable of fathering children must agree to use an effective method of contraception for the duration of the trial.
* Subjects on bisphosphonate therapy must be on a stable dose and must have started therapy > 4 weeks prior to protocol therapy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Use of red blood cell or platelet transfusions within 4 weeks of treatment
* Use of hematopoietic growth factors within 4 weeks of treatment
* Prior cytotoxic chemotherapy and/or radiation therapy within 4 weeks of treatment
* Prior radiation therapy encompassing >25% of skeleton (see Appendix C)
* Prior treatment with 89Strontium or 153Samarium containing compounds (e.g. Metastron®, Quadramet®)
* Platelet count <150,000/mm3 or known primary qualitative platelet disorder
* Absolute neutrophil count (ANC) <2,000/mm3
* Hematocrit <30 percent and Hemoglobin < 10 g/dL
* Abnormal coagulation profile (PT or INR, PTT > 1.3x ULN) unless on therapeutic anticoagulation - see concomitant meds section
* Serum creatinine >2.5 mg/dL
* AST (SGOT) >2x ULN
* Bilirubin (total) >1.5x ULN; subjects with Gilbert's syndrome will be allowed if direct bilirubin is within institutional normal limits
* Active serious infection
* Active angina pectoris or NY Heart Association Class III-IV
* ECOG Performance Status > 2
* Life expectancy <12 months
* History of deep vein thrombosis and/or pulmonary embolus within 1 month of study entry
* Other serious illness(es) involving the cardiac, respiratory, CNS, renal, hepatic or hematological organ systems which might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study
* Prior investigational therapy (medications or devices) within 4 weeks of treatment. Furthermore, other investigational therapy is not permitted during the treatment phase.
* Prior use of ketoconazole for the purposes of prostate cancer therapy for greater than 1 month
* Known history of HIV. The effects of J591 are unknown in this population. Furthermore, ketoconazole has many well-described drug-drug interactions which could affect antiviral therapy. If necessary, this population will be studied separately.
* Currently active other malignancy other than non-melanoma skin cancer. Patients are considered not to have "currently active" malignancy if they have completed any necessary therapy and are considered by their physician to be at less than 30% risk of relapse.

  - Known history of known myelodysplastic syndrome
* Adrenal hormone inhibitors (other than ketoconazole) within 4 weeks prior to study enrollment
* Finasteride (Propecia® or Proscar®) or dutasteride (Avodart®) within 4 weeks of enrollment
* Patients on corticosteroids prior to enrollment must have either discontinued and shown biochemical progression or have biochemical progression on a stable dose

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2026-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Scott T Tagawa, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (9):
- United States (9):
  - Cedars Sinai, Los Angeles, California
  - USC/Norris Comprehensive cancer center, Los Angeles, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Weill Cornell Medical College, New York, New York
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 1. 177Lu-J591+Ketoconzole: Ketoconazole 400 mg 3 times a day plus hydrocortisone 20 mg AM, 10 mg PM x 4 weeks followed by 177Lu-J591 Infusion, continue ketoconazole and hydrocortisone
  177Lu-J591: 177Lu-J591 70 mCi/m2 on day 29 (+/- 2 days) of treatment
  Ketoconazole: Ketoconazole at a dose of 400 mg (two 200 mg tabs) to be taken orally (preferably on an empty stomach) three times per day (total daily dose of 1200 mg)
  Hydrocortisone: Hydrocortisone at a dose of 20 mg orally each morning, 10 mg orally each evening (total daily dose of 30 mg)
Period: Overall Study
Arm/Group | 1. 177Lu-J591+Ketoconzole | 2. 111In-J591 + Ketoconazole
Started | 38 | 17
Completed | 38 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1. 177Lu-J591+Ketoconzole | 2. 111In-J591 + Ketoconazole | Total
Number analyzed (Participants) | 38 | 17 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 5 | 16
  >=65 years | 27 | 12 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 38 | 17 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 38 | 14 | 52
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 34 | 15 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 38 | 17 | 55

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Free of Radiographically Evident Metastases From Baseline to 18 Months After Study Drug Administration
Description: Subjects will perform a CT and/or MRI scan of the abdomen and pelvis, chest x-ray or CT scan of the chest and bone scan to determine the proportion of participants free of radiographically evident metastases from baseline to 18 months after study drug administration.
Time Frame: Baseline and 18 months after study drug administration
Measure: Number; unit: proportion of participants
Arm/Group | 1. 177Lu-J591+Ketoconzole | 2. 111In-J591 + Ketoconazole
Number analyzed (Participants) | 38 | 17
proportion of participants | 0.50 | 0.24
Statistical Analysis 1: Comparison: 1. 177Lu-J591+Ketoconzole vs 2. 111In-J591 + Ketoconazole; Test type: Superiority; p = 0.08, Fisher Exact; proportion difference = 0.26, 95% CI 2-sided [0.008 to 0.52] — Direction = 177Lu-J591 + Ketoconazole proportion free of radiographically evident metastases minus 111ln-J591 + Ketoconazole proportion free of radiographically evident metastases

2. Secondary Outcome: Change in PSA Response Rate
Description: PSA response will be determined by comparing the PSA levels after therapy to the baseline and pre-treatment PSA via blood specimens
Time Frame: Collected at screening, V2, V3, V5, V9 then every 4 weeks till PSA progression or end of study at approximately 100 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 years
Arm/Group | 1. 177Lu-J591+Ketoconzole | 2. 111In-J591 + Ketoconazole
All-Cause Mortality (participants affected / at risk) | 13/38 | 5/17
Serious Adverse Events (participants affected / at risk) | 2/38 | 0/17
Other Adverse Events (participants affected / at risk) | 36/38 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. 177Lu-J591+Ketoconzole (N=38) | 2. 111In-J591 + Ketoconazole (N=17)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1. 177Lu-J591+Ketoconzole (N=38) | 2. 111In-J591 + Ketoconazole (N=17)
Infection (Gastrointestinal disorders) | 6 | 4
ALT Increase (Blood and lymphatic system disorders) | 5 | 6
Anemia (Blood and lymphatic system disorders) | 21 | 8
Anorexia (Metabolism and nutrition disorders) | 9 | 2
Any Pain (General disorders) | 18 | 7
AST Increase (Blood and lymphatic system disorders) | 6 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 9
Bilirubin Increase (Hepatobiliary disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 8 | 3
Creatinine Increase (Investigations) | 6 | 4
Depression (Psychiatric disorders) | 5 | 3
Diarrhea (Gastrointestinal disorders) | 6 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Edema in Limbs (Musculoskeletal and connective tissue disorders) | 8 | 4
Fatigue (General disorders) | 21 | 10
Headaches (Nervous system disorders) | 6 | 2
Hematuria (Renal and urinary disorders) | 4 | 1
Hypokalemia (Metabolism and nutrition disorders) | 5 | 0
Insomnia (Psychiatric disorders) | 11 | 2
Lymphocyte Count Decreased (Investigations) | 9 | 1
Neutropenia (Blood and lymphatic system disorders) | 19 | 2
Pain in Extremities (Musculoskeletal and connective tissue disorders) | 10 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 26 | 3
Vomiting (Gastrointestinal disorders) | 4 | 2
WBC Decreased (Investigations) | 10 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT00859781/Prot_SAP_000.pdf